CLINICAL TRIAL: NCT06352840
Title: Novel Web-based, Self-directed Intervention for Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sara Till, MD, MPH, Assistant Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00231526; 5K23HD099283-03 (NIH)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pelvic Pain; Endometriosis
Keywords: Quality of life; Cognitive Behavioral Therapy
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and outcome assessors will be blinded to study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monitoring progress plus usual care (Other): Participants will have access to the monitoring progress web-based symptom monitoring program.
  Interventions: Behavioral: Control Group website
- My Pelvic Plan plus usual care (Experimental): Participants will have access to My Pelvic Plan program.
  Interventions: Behavioral: My Pelvic Plan Website

INTERVENTIONS:
Behavioral: My Pelvic Plan Website — This is a self-directed program which integrates patient education about conditions that frequently contribute to pelvic pain, as well as instruction on cognitive and behavioral restructuring, self-administration of acupressure, engaging in physical activity, and a brief introduction to pelvic floor physical therapy techniques. Participants will have open access to the program over the 6-month intervention period. The intervention will be comprised of an active (12-week) phase and a maintenance (3-month) phase. Participants will receive a weekly text or email prompt directing patients to a specific module. All participants will receive prompts to the same modules for the first four weeks of the study, then during the next 8 weeks, participants will receive prompts to modules that corresponded to the most impactful symptoms on participant's baseline questionnaires. Following 12-week active phase, all participants will enter the maintenance phase.
  Arms: My Pelvic Plan plus usual care
Behavioral: Control Group website — Patients in the control group will undergo an active control intervention in which participants receive open access to a separate website that contains only the Monitoring Progress symptom tracker subpage over the 6-month study period. Control group participation will also be divided into an active (12-week) phase and a maintenance (3-month) phase. Similar to the intervention group, the control group will receive a weekly text (first 12 weeks) or email prompt directing them to a specific module or portion of the respective website. During the maintenance phase of the study, participants will receive monthly prompts to the Monitoring Progress subpage (without prompting to a specific symptom or activity).
  Arms: Monitoring progress plus usual care

SUMMARY:
The study is being completed to evaluate the effectiveness of a web-based, self-management program for patients with Chronic Pelvic Pain (CPP).

The overall hypothesis is that patients with chronic pelvic pain that have access to the My Pelvic Plan program will demonstrate improvements in pain, physical function, and quality of life with this integrative self-management approach.

ELIGIBILITY:
Inclusion Criteria:

* Participants have chronic pelvic pain, defined by the protocol for ≥ 6-month duration, and is non-cyclic, occurring for at least 14 days of each month.
* Must be currently receiving care within Department of Obstetrics and Gynecology at the University of Michigan for treatment of chronic pelvic pain
* Access to internet via computer or smartphone
* English-language proficiency (current version of the website is in English)

Exclusion Criteria:

* Underwent gynecologic surgery within 3 months of screening visit
* Plan to undergo gynecologic surgery within 6 months following screening visit
* Pregnant (self-reported) at time of screening visit. Will not exclude patients that become pregnant during the course of the study.
* Severe physical impairment precluding participating in internet-based program (for example, complete blindness or deafness)
* Current psychiatric disorder with history of psychosis (for example, schizophrenia, schizoaffective disorder, delusional disorder),
* Current suicidal ideation or suicide attempt within 2 years of screening visit. The study will screen for severe depression and suicidality at each questionnaire time point and have developed a robust triage and referral plan.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman (female sex assigned at birth, may include cis-gender, trans-gender, nonbinary)
Enrollment: 69 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference short form (SF) 4a between groups | 3 months
  There are four questions that participants will answer from not at all (1) - very much (5). Scores range from 4-20, with higher scores meaning more interference.
PROMIS pain intensity 1a between groups | 3 months
  There is one question that participants will answer no pain (0) - worst pain (10). Lower score means less pain.
PROMIS Self Efficacy for Managing Symptoms SF 4a between groups | 3 months
  There are four questions that participants will answer from I am not all confident (1) - I am very confident (5). Scores range from 4-20, with higher scores meaning more confident.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference short form (SF) 4a between groups | 6 months
  There are four questions that participants will answer from not at all (1) - very much (5). Scores range from 4-20, with higher scores meaning more interference.
PROMIS pain intensity 1a between groups | 6 months
  There is one question that participants will answer no pain (0) - worst pain (10). Lower score means less pain.
PROMIS Self Efficacy for Managing Symptoms SF 4a between groups | 6 months
  There are four questions that participants will answer from I am not all confident (1) - I am very confident (5). Scores range from 4-20, with higher scores meaning more confident.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Till, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No